CLINICAL TRIAL: NCT01978470
Title: External Trigeminal Nerve Stimulation for Epilepsy
Brief Title: External Trigeminal Nerve Stimulation for Drug Resistent Epilepsy
Acronym: eTNS for DRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeuroSigma, Inc. (Industry)
Collaborators: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NS-076014-01; NCT01607567 (obsolete NCT alias)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Seizure Disorder
Keywords: epilepsy; drug resistent epilepsy; partial onset seizures; trigeminal nerve stimulation; neuromodulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active (Experimental): Trigeminal nerve stimulation
  Interventions: Device: External Trigeminal Nerve Stimulation (eTNS)

INTERVENTIONS:
Device: External Trigeminal Nerve Stimulation (eTNS) — External stimulation of the trigeminal nerve.
  Other Names: eTNS

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of the NeuroSigma eTNS system.

DETAILED DESCRIPTION:
This study evaluates the safety and tolerability of the NeuroSigma eTNS system for the treatment of drug resistent partial seizures.

Up to 20 subjects, ages 18 - 75, with partial epilepsy will be enrolled in an acute 4-week tolerability study at Olive View/UCLA Medical Center .......

Enrolled subjects will be asked to maintain an accurate seizure calendar, and will be seen at the initial visit, then at two and four weeks.......

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Partial onset seizures (complex partial or secondary generalized tonic-clonic)
* At least one seizure every three months
* No serious or progressive medical or psychiatric illness
* At least one complex partial or generalized tonic-clonic seizure in the last three months
* MRI or EEG consistent with localization-related or partial epilepsy
* Exposure to at least two anti-epileptic drugs at adequate doses
* Concurrent use of at least one anti-epileptic drug at adequate doses
* No change in anti-epileptic drug dose for at least 30 days prior to study enrollment

Exclusion Criteria:

* Vagus nerve stimulation (VNS)
* History of non-epileptic seizures
* Inability to maintain accurate seizure calendars (self or caregiver)
* Frequent use of benzodiazepines for seizure clusters defined as greater that four times per month
* History of facial pain or trigeminal neuralgia
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Safety of eTNS | Four weeks
  Number and percent of subjects with adverse events related to the device at four weeks.

SECONDARY OUTCOMES:
Beck Depression Inventory | Four weeks
  Percentage change in Beck Depression Inventory score at four weeks compared to initial visit.
Quality of Life | Four weeks
  Absolute change in QOLIE-31 (Quality of Life in Epilepsy) Inventory scale and sub-scales at four weeks.
Systolic Blood Pressure and Heart Rate | Four weeks
  Absolute and percent change in systolic blood pressure and heart rate at four weeks compared to initial visit.
Skin Irritation | Four weeks
  Number and percentage of subjects with skin irritation > 1 on a standardized scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View/UCLA Medical Center, Sylmar, California, United States